CLINICAL TRIAL: NCT07364045
Title: Mechanisms Mediating Reversible Lipotoxicity of the Pancreas in Obesity-induced Type 2 Diabetes: Edinburgh Diabetes Remission Study (EDRS)
Brief Title: Pancreas Lipotoxicity in T2D: Edinburgh Diabetes Remission Study (EDRS)
Acronym: EDRS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC23027
Record Dates: First submitted 2026-01-08; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Obesity; Remission; Weight loss
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Weight Loss | interventions — Thymidine; Caloric Restriction

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of four parallel groups based on baseline glycemic status: non-diabetic, pre-diabetic, short-duration type 2 diabetes (<6 years), and long-duration type 2 diabetes (>10 years). All groups receive the same dietary intervention (8-12-week Total Diet Replacement followed by food reintroduction and weight maintenance), but remain in their respective groups for analysis. No crossover or sequential assignment occurs.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Non-Diabetic Group (Experimental): Participants without diabetes who are overweight or obese (BMI 30-45 kg/m²) will undergo an 8-12-week Total Diet Replacement (TDR) intervention (~800 kcal/day) followed by food reintroduction and weight maintenance. Includes metabolic testing, MRI scans, and blood sampling at baseline and follow-up.
  Interventions: Behavioral: Total Diet Replacement (TDR) Program
- Pre-Diabetic Group (Experimental): Participants with pre-diabetes who are overweight or obese (BMI 30-45 kg/m²) will receive the same TDR intervention and follow-up schedule as the Non-Diabetic Group, with additional oral glucose tolerance testing during screening.
  Interventions: Behavioral: Total Diet Replacement (TDR) Program
- Short-Duration Type 2 Diabetes Group (Experimental): Participants with type 2 diabetes diagnosed <6 years who are overweight or obese (BMI 30-45 kg/m²) will undergo the TDR intervention and extended follow-up (up to 12-24 months) with additional metabolic visits and blood sampling.
  Interventions: Behavioral: Total Diet Replacement (TDR) Program
- Long-Duration Type 2 Diabetes Group (Experimental): Participants with type 2 diabetes diagnosed >10 years who are overweight or obese (BMI 30-45 kg/m²) will receive the same TDR intervention and standard follow-up schedule as other arms.
  Interventions: Behavioral: Total Diet Replacement (TDR) Program

INTERVENTIONS:
Behavioral: Total Diet Replacement (TDR) Program — Participants will follow a structured Total Diet Replacement (TDR) program consisting of approximately 800 kcal/day using commercially available soups and shakes for 8-12 weeks. This is followed by a 2-week food reintroduction phase and a weight maintenance phase up to 6 months, supervised by a research dietitian. The intervention aims to induce rapid weight loss and assess its impact on intrapancreatic fat, insulin secretion, and type 2 diabetes remission. All participants receive dietary counseling and monitoring throughout the study.
  Other Names: Low-Calorie Diet; Meal Replacement Program

SUMMARY:
This study aims to investigate how fat accumulation in the pancreas contributes to the development of type 2 diabetes (T2D), and how weight loss may reverse this process. Previous research has shown that reducing body weight can lead to diabetes remission, and this was accompanied by lowering intrapancreatic fat and restoration of insulin secretion, but the mechanisms behind this are not fully understood. In particular, the study aims to unravel the role of hepatic de novo lipogenesis (DNL) and lipoprotein metabolism on pancreas lipotoxicity and beta cell recovery after weight loss.

Four groups of participants will be recruited (n=26 per group): non-diabetic, pre-diabetic, short-duration T2D (<6 years), and long-duration T2D (>10 years). Participants will be aged between 45 and 79 years and have a BMI between 30 and 45 kg/m². All participants will follow a structured weight loss programme using an 800 kcal/day Total Diet Replacement (TDR) for 8-12 weeks, followed by dietary support to maintain weight loss. The study is sponsored by NHS-Lothian and the University of Edinburgh and will be carried out at the Clinical Research Facility, Royal infirmary of Edinburgh by a specialist team (Senior Diabetes Research Nurse, Clinical Fellow, and Research Dietitian).

The primary endpoint of this study is to achieve a 10-15% reduction in body weight (~10 kg) through a low-calorie diet (800 kcal/day) to induce T2D remission and maintain this weight loss with structured dietary support for up to 6-12 months. The primary aim is to compare hepatic de novo lipogenesis-the conversion of sugar into fat by the liver-and lipoprotein export among the groups, and to examine how these parameters change in response to weight loss, improvement in metabolic status, and restoration of normal pancreatic function.

Secondary endpoints include changes in weight, HbA1c, intraorgan fat (liver/pancreas), pancreas volume and tissue characteristics, beta cell mass and function (MRI/mixed meal test), circulating blood markers (i.e. lipids, exosomes, adipokines, and inflammatory markers), and the change in adipose tissue biology (fat biopsies).

Ultimately, this study aims to understand the mechanisms of T2D remission. It will help clarify the sequence of metabolic events leading to reversible pancreatic lipotoxicity and may inform the development of new, targeted therapies for T2D.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese (BMI: 30-45 kg/m²) who have had T2D for less than 6 years or longer than 10 years, and are on treatment with diet alone or diet plus oral medication.
* Overweight/obese (BMI: 30-45 kg/m²) who are at pre-diabetes stage, defined as fasting blood glucose 5.6-6.9 mmol/L.
* Overweight/obese (BMI: 30-45 kg/m²) who are non-diabetic (control group).
* Age between 45 and 79 years inclusive.
* Post-menopausal women only (to exclude sex hormone effects on lipid metabolism).
* Good communication in English (able to give informed consent and follow dietary advice).
* Willing and able to adhere to the study protocol, including dietary intervention and scheduled follow-up visits.

Exclusion Criteria:

* Insulin therapy
* HbA1c >12% (108 mmol/mol)
* Weight loss >5 kg in last 6 months
* Recent MI (within 6 months)
* Known cancer in last 5 years
* First-degree relatives of people with T2D (control group)
* History of gestational diabetes
* MRI contraindications (metal implants, claustrophobia)
* Alcohol >14 units/week
* Advanced kidney or liver disease
* Use of steroids or antipsychotics
* Participation in another clinical trial
* Life expectancy <1 year
* Allergy to local anaesthetic (for biopsy subgroup)
* Any disorder that may jeopardise safety or compliance

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in body weight from baseline to 6-12 months post-intervention | Baseline, 6 months, and 12 months post-intervention
  The primary endpoint is achieving a 10-15% reduction in body weight (~10 kg) through a low-calorie diet (800 kcal/day) to induce T2D remission and maintain this weight loss with structured dietary support for up to 6-12 months. The study will also compare four participant groups (non-diabetic, pre-diabetic, short-duration T2D, long-duration T2D) in terms of hepatic de novo lipogenesis and lipoprotein export, and examine changes in these parameters in response to weight loss and improved metabolic status.
Change in hepatic de novo lipogenesis measured using stable isotope tracers | Baseline, 6 months, and 12 months
  Hepatic de novo lipogenesis will be quantified using stable isotope tracer methodology (deuterated water) at baseline and after intervention.

SECONDARY OUTCOMES:
Change in liver and pancreas fat measured by MRI | Baseline, 6 months, and 12 months
  Hepatic and intrapancreatic fat will be assessed by MRI at baseline and after intervention to evaluate the effect of weight loss on intraorgan fat deposition.
Change in beta-cell function assessed by C-peptide response during mixed meal test | Baseline, 6 months, and 12 months
  Beta-cell function will be evaluated using C-peptide modeling during a standardised mixed meal test at baseline and after intervention.
Change in circulating lipoproteins and lipids | Baseline, 6 months, and 12 months
  Lipoproteins (i.e. VLDL) and plasma/serum lipids will be measured using ultracentrifugation and mass spectrometry techniques.
Change in pancreas morphology and tissue inflammation | Baseline, 6 months, and 12 months
  Pancreas size, shape, and tissue inflammation will be evaluated by assessed by MR methods at baseline and after intervention.
Change in adipose tissue biology | Baseline and 6 months post-intervention
  MRI will be used to assess fat saturation, and fat biopsies will be performed to evaluate molecular changes in adipose tissue biology.
Change in circulating markers | Baseline and 6 months post-intervention
  Changes in circulating adipokines, inflammatory markers, and exosomes will be measured using commercial kits to assess systemic metabolic responses to weight loss.
Change in lipid profile | Baseline, 6 months, and 12 months
  Fasting lipids (TGs, HDL, LD cholesterol) will be measured at baseline and after intervention at NHS- accredited lab to assess cardiometabolic improvement.
Change in blood pressure | Baseline, 6 months, and 12 months
  Blood pressure will be measured at baseline and after intervention to assess cardiometabolic improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Al-Mrabeh, PhD, Principal Investigator — University of Edinburgh
Locations (1):
- Clinical Research Facility, Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided